CLINICAL TRIAL: NCT02362594
Title: Adjuvant Immunotherapy With Anti-PD-1 Monoclonal Antibody Pembrolizumab (MK-3475) Versus Placebo After Complete Resection of High-risk Stage III Melanoma: A Randomized, Double- Blind Phase 3 Trial of the EORTC Melanoma Group
Brief Title: Study of Pembrolizumab (MK-3475) Versus Placebo After Complete Resection of High-Risk Stage III Melanoma (MK-3475-054/1325-MG/KEYNOTE-054)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: European Organisation for Research and Treatment of Cancer (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-054; 1325-MG (Other: European Organisation for Research and Treatment of Cancer); 163277 (Registry Identifier: JAPIC-CTI); KEYNOTE-054 (Other: MSD); MK-3475-054 (Other: MSD); 2023-509136-25-00 (Registry Identifier: EU CT); U1111-1309-6016 (Registry Identifier: UTN); 2014-004944-37 (EudraCT Number)
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Melanoma
Keywords: Programmed Cell Death-1 (PD-1); Programmed Cell Death 1 (PD1); Programmed Cell Death-Ligand 1 (PD-L1, PDL1); Programmed Cell Death-Ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab (Experimental): In Part 1, participants receive pembrolizumab 200 mg intravenously (IV) as post-surgery therapy every 3 weeks (Q3W) for up to 1 year. During Part 2, participants with documented recurrence may receive optional re-treatment with pembrolizumab Q3W for up to 2 years or disease progression.
  Interventions: Biological: pembrolizumab
- Placebo (Placebo Comparator): In Part 1, participants receive placebo IV as post-surgery therapy Q3W. During Part 2, participants with documented recurrence who received placebo in Part 1 may receive optional treatment with pembrolizumab Q3W for up to 2 years or disease progression.
  Interventions: Drug: placebo

INTERVENTIONS:
Biological: pembrolizumab — Pembrolizumab 200 mg administered intravenously (IV) on Day 1 of each 21-day cycle
  Other Names: KEYTRUDA®; MK-3475; SCH 900475
  Arms: Pembrolizumab
Drug: placebo — Normal saline solution administered IV on Day 1 of each 21-day cycle
  Arms: Placebo

SUMMARY:
This study will assess whether post-surgery therapy with pembrolizumab improves recurrence-free survival (RFS) as compared to placebo for high-risk participants with melanoma (Stage IIIA [> 1 mm metastasis], IIIB and IIIC). The study will also assess whether pembrolizumab improves RFS versus placebo in the subgroup of participants with programmed cell death-ligand 1 (PD-L1)-positive tumor expression. Participants will be stratified for stage of disease and region and then will be randomly assigned to receive either pembrolizumab or placebo as post-surgery therapy in Part 1. In Part 2, participants who experience a disease recurrence are eligible for pembrolizumab treatment (if treated with placebo in Part 1) or pembrolizumab rechallenge (if treated with pembrolizumab in Part 1).

DETAILED DESCRIPTION:
As of Amendment 8, enrollment in Part 2 has closed, and an optional pembrolizumab extension study will not be available to participants after study closure.

ELIGIBILITY:
Inclusion criteria:

* Completely resected Stage III melanoma
* Tumor tissue available for evaluation of PD-L1 expression
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* No prior therapy for melanoma except surgery for primary melanoma lesions (or previously treated with interferon for thick primary melanomas without evidence of lymph node involvement are eligible)
* Female participants of childbearing potential should be willing to use adequate methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication
* Male participants should agree to use an adequate method of birth control starting with the first dose of study therapy through 120 days after the last dose of study medication

Exclusion criteria:

* Mucosal or ocular melanoma
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis
* History of or current interstitial lung disease
* History of hematologic or primary solid tumor malignancy, unless no evidence of that disease for 5 years
* Active autoimmune disease that has required systemic treatment in past 2 years
* Active infection requiring therapy
* Unstable hyperthyroidism or hypothyroidism
* Diagnosis of immunodeficiency
* Systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study medication
* Known history of human immunodeficiency virus (HIV), active Hepatitis B or C
* Treatment with live vaccine within 30 days prior to the first dose of study medication are not eligible
* Prior treatment with any anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA4) monoclonal antibody or anti-programmed cell death receptor 1 (PD-1), anti-programmed cell death receptor ligand 1 (PD-L1), or anti-programmed cell death receptor ligand 2 (PD-L2) agent, or prior participation in any Merck pembrolizumab clinical trial
* Currently participating and receiving study therapy, or participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of study medication
* Pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of study medication
* Participant is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or Sponsor staff directly involved with this trial without prospective Institutional Review Board approval (by chair or designee) is given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2015-07-16 (Actual); Primary Completion 2018-01-08 (Actual); Study Completion 2026-11-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Buhrer E, Kicinski M, Mandala M, Pe M, Long GV, Atkinson V, Blank CU, Haydon A, Dalle S, Khattak A, Carlino MS, Meshcheryakov A, Sandhu S, Puig S, Schadendorf D, Jamal R, Rutkowski P, van den Eertwegh AJM, Coens C, Grebennik D, Krepler C, Robert C, Eggermont AMM. Adjuvant pembrolizumab versus placebo in resected stage III melanoma (EORTC 1325-MG/KEYNOTE-054): long-term, health-related quality-of-life results from a double-blind, randomised, controlled, phase 3 trial. Lancet Oncol. 2024 Sep;25(9):1202-1212. doi: 10.1016/S1470-2045(24)00338-3. Epub 2024 Aug 12. PMID 39146951
- [Derived] Eggermont AMM, Kicinski M, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Meshcheryakov A, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Boers-Sonderen M, Di Giacomo AM, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, van Akkooi ACJ, Lorigan P, Grebennik D, Krepler C, Marreaud S, Suciu S, Robert C. Five-Year Analysis of Adjuvant Pembrolizumab or Placebo in Stage III Melanoma. NEJM Evid. 2022 Nov;1(11):EVIDoa2200214. doi: 10.1056/EVIDoa2200214. Epub 2022 Sep 10. PMID 38319852
- [Derived] Kennedy OJ, Kicinski M, Valpione S, Gandini S, Suciu S, Blank CU, Long GV, Atkinson VG, Dalle S, Haydon AM, Meshcheryakov A, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Di Giacomo AM, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, van Akkooi ACJ, Robert C, Eggermont AMM, Lorigan P, Mandala M. Prognostic and predictive value of beta-blockers in the EORTC 1325/KEYNOTE-054 phase III trial of pembrolizumab versus placebo in resected high-risk stage III melanoma. Eur J Cancer. 2022 Apr;165:97-112. doi: 10.1016/j.ejca.2022.01.017. Epub 2022 Feb 24. PMID 35220182
- [Derived] Bottomley A, Coens C, Mierzynska J, Blank CU, Mandala M, Long GV, Atkinson VG, Dalle S, Haydon AM, Meshcheryakov A, Khattak A, Carlino MS, Sandhu S, Puig S, Ascierto PA, Larkin J, Lorigan PC, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Di Giacomo AM, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, van Akkooi ACJ, Krepler C, Ibrahim N, Marreaud S, Kicinski M, Suciu S, Robert C, Eggermont AMM; EORTC Melanoma Group. Adjuvant pembrolizumab versus placebo in resected stage III melanoma (EORTC 1325-MG/KEYNOTE-054): health-related quality-of-life results from a double-blind, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 May;22(5):655-664. doi: 10.1016/S1470-2045(21)00081-4. Epub 2021 Apr 12. PMID 33857414
- [Derived] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson VG, Dalle S, Haydon AM, Meshcheryakov A, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Di Giacomo AM, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan PC, van Akkooi ACJ, Krepler C, Ibrahim N, Marreaud S, Kicinski M, Suciu S, Robert C; EORTC Melanoma Group. Adjuvant pembrolizumab versus placebo in resected stage III melanoma (EORTC 1325-MG/KEYNOTE-054): distant metastasis-free survival results from a double-blind, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 May;22(5):643-654. doi: 10.1016/S1470-2045(21)00065-6. Epub 2021 Apr 12. PMID 33857412
- [Derived] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson VG, Dalle S, Haydon AM, Meshcheryakov A, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Di Giacomo AM, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan PC, van Akkooi ACJ, Krepler C, Ibrahim N, Marreaud S, Kicinski M, Suciu S, Robert C. Longer Follow-Up Confirms Recurrence-Free Survival Benefit of Adjuvant Pembrolizumab in High-Risk Stage III Melanoma: Updated Results From the EORTC 1325-MG/KEYNOTE-054 Trial. J Clin Oncol. 2020 Nov 20;38(33):3925-3936. doi: 10.1200/JCO.20.02110. Epub 2020 Sep 18. PMID 32946353
- [Derived] Eggermont AMM, Kicinski M, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Di Giacomo AM, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan PC, Krepler C, Ibrahim N, Marreaud S, van Akkooi A, Robert C, Suciu S. Association Between Immune-Related Adverse Events and Recurrence-Free Survival Among Patients With Stage III Melanoma Randomized to Receive Pembrolizumab or Placebo: A Secondary Analysis of a Randomized Clinical Trial. JAMA Oncol. 2020 Apr 1;6(4):519-527. doi: 10.1001/jamaoncol.2019.5570. PMID 31895407
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Eggermont AMM, Blank CU, Mandala M, Long GV, Atkinson V, Dalle S, Haydon A, Lichinitser M, Khattak A, Carlino MS, Sandhu S, Larkin J, Puig S, Ascierto PA, Rutkowski P, Schadendorf D, Koornstra R, Hernandez-Aya L, Maio M, van den Eertwegh AJM, Grob JJ, Gutzmer R, Jamal R, Lorigan P, Ibrahim N, Marreaud S, van Akkooi ACJ, Suciu S, Robert C. Adjuvant Pembrolizumab versus Placebo in Resected Stage III Melanoma. N Engl J Med. 2018 May 10;378(19):1789-1801. doi: 10.1056/NEJMoa1802357. Epub 2018 Apr 15. PMID 29658430
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As of the 02-Oct-2017 interim database cut-off date, of the 1019 randomized participants in Part 1, 544 had completed Part 1 and 62 were continuing in Part 1. This interim results disclosure is for Part 1 only.
Groups:
- Pembrolizumab: In Part 1, participants received pembrolizumab 200 mg intravenously (IV) as post-surgery therapy every 3 weeks (Q3W) for up to 1 year.
- Placebo: In Part 1, participants received placebo IV as post-surgery therapy Q3W.
Period: Overall Study
Arm/Group | Pembrolizumab | Placebo
Started | 514 | 505
Treated | 509 | 502
Continuing Part 1 Adjuvant Therapy | 41 | 21
Completed (Completed Part 1 Adjuvant Therapy) | 264 | 280
Not Completed | 250 | 225

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: In Part 1, participants received pembrolizumab 200 mg IV as post-surgery therapy Q3W for up to 1 year.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Placebo | Total
Number analyzed (Participants) | 514 | 505 | 1019
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (13.6) | 53.7 (14.2) | 53.8 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 201 | 391
  Male | 324 | 304 | 628
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Programmed Death-Ligand 1 (PD-L1) Tumor Status [Count of Participants; unit: Participants] — Tumor PD-L1 status was assessed by immunohistochemistry (IHC) and recorded as positive (≥1% PD-L1 IHC), negative (<1% PD-L1 IHC), or undetermined level of expression (indeterminate PD-L1 IHC).
  Participants
    PD-L1 Positive | 428 | 425 | 853
    PD-L1 Negative | 59 | 57 | 116
    Undetermined | 27 | 23 | 50
Melanoma Stage [Count of Participants; unit: Participants] — Participants were stratified by melanoma stage using the American Joint Committee on Cancer (AJCC) 7th edition stage as follows: Stage IIIA (with >1 mm metastasis), Stage IIIB, Stage IIIC with 1-3 positive lymph nodes (LN+), and Stage IIIC with ≥4 LN+.
  Participants
    Stage IIIA (> 1 mm) | 80 | 80 | 160
    Stage IIIB | 237 | 230 | 467
    Stage IIIC (1-3 LN+) | 95 | 93 | 188
    Stage IIIC (≥4 LN+) | 102 | 102 | 204
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 38 | 37 | 75
  Europe | 341 | 336 | 677
  Australia/New Zealand | 111 | 112 | 223
  Other | 24 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants With Recurrence-Free Survival (RFS) At 6 Months Among All Participants
Description: RFS was defined as the time between the date of randomization and the date of first melanoma recurrence (local, regional, distant metastasis) or death (whatever the cause), whichever occurred first. For participants who remained alive and whose disease had not recurred, RFS was censored on the date of last visit/contact with disease assessments. The percentage of participants with RFS at Month 6 was reported for all participants in both treatment arms of Part 1.
Time Frame: 6 months
Population: All randomized participants in Part 1.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 514 | 505
Percentage of Participants | 82.2 [78.6 to 85.3] | 73.3 [69.2 to 77.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Comparison of RFS time-to-event distribution between the 2 treatment arms was based on Cox regression model with treatment as a covariate stratified by stage (IIIA [>1 mm metastasis] vs. IIIB vs. IIIC 1-3 nodes vs. IIIC ≥4 nodes) as indicated at randomization; Test type: Superiority; p < 0.0001, Regression, Cox — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.57, 98.4% CI 2-sided [0.43 to 0.74]

2. Primary Outcome: Part 1: Percentage of Participants With Recurrence-Free Survival (RFS) At 6 Months Among Participants With PD-L1-positive Tumor Expression
Description: RFS was defined as the time between the date of randomization and the date of first melanoma recurrence (local, regional, distant metastasis) or death (whatever the cause), whichever occurred first. For participants who remained alive and whose disease had not recurred, RFS was censored on the date of last visit/contact with disease assessments. The percentage of participants with RFS at Month 6 was reported for all participants with PD-L1-positive tumors in both treatment arms of Part 1.
Time Frame: 6 months
Population: All randomized participants in Part 1 with PD-L1-positive tumors.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 428 | 425
Percentage of Participants | 83.8 [80.0 to 87.0] | 75.4 [71.0 to 79.2]
Statistical Analysis 1: Comparison: Pembrolizumab vs Placebo; Comparison of RFS time-to-event distribution between the 2 treatment arms (PD-L1-positive participants) was based on Cox regression model with treatment as a covariate stratified by stage (IIIA [>1 mm metastasis] vs. IIIB vs. IIIC 1-3 nodes vs. IIIC ≥4 nodes) as indicated at randomization; Test type: Superiority; p < 0.0001, Regression, Cox — One-sided p-value based on log-rank test; Hazard Ratio (HR) = 0.54, 95.0% CI 2-sided [0.42 to 0.69]

3. Secondary Outcome: Distant Metastases-free Survival (DMFS) in All Participants
Description: DMFS will be defined as the time between the date of randomization and the date of first distant metastasis or date of death (whatever the cause), whichever occurs first. For participants who remain alive and distant metastasis-free, DMFS will be censored on the date of last visit/contact with disease assessments. The percentage of participants with DMFS will be reported for all participants in both treatment arms.
Time Frame: Up to approximately 11 years
Reporting Status: Not Posted, anticipated posting 2026-11

4. Secondary Outcome: Distant Metastases-free Survival (DMFS) for Participants With PD-L1-positive Tumor Expression
Description: Description:
  DMFS will be defined as the time between the date of randomization and the date of first distant metastasis or date of death (whatever the cause), whichever occurs first. For participants who remain alive and distant metastasis-free, DMFS will be censored on the date of last visit/contact with disease assessments. The percentage of participants with DMFS will be reported for all participants with PD-L1-positive tumors in both treatment arms.
Time Frame: Up to approximately 11 years
Reporting Status: Not Posted, anticipated posting 2026-11

5. Secondary Outcome: Overall Survival (OS) for All Participants
Description: OS will be defined as the time from the date of randomization to the date of death, whatever the cause. The follow-up of participants still alive will be censored at the moment of last visit/contact. OS will be reported for all participants in both treatment arms.
Time Frame: Up to approximately 11 years
Reporting Status: Not Posted, anticipated posting 2026-11

6. Secondary Outcome: Overall Survival (OS) for Participants With PD-L1-positive Tumor Expression
Description: OS will be defined as the time from the date of randomization to the date of death, whatever the cause. The follow-up of participants still alive will be censored at the moment of last visit/contact. OS will be reported for all participants with PD-L1-positive tumors in both treatment arms.
Time Frame: Up to approximately 11 years
Reporting Status: Not Posted, anticipated posting 2026-11

7. Secondary Outcome: Number of Participants Who Experienced At Least 1 Adverse Event (AE)
Description: An AE is defined as "any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with this treatment". An AE can therefore be any unfavorable and unintended signs (such as rash or enlarged liver), symptoms (such as nausea or chest pain), an abnormal laboratory finding (including results of blood tests, x-rays or scans) or a disease temporarily associated with the use of the protocol treatment, whether or not considered related to the investigational medicinal product. The number of participants who experienced at least 1 AE was reported for all participants in each treatment arm.
Time Frame: Up to 22 months
Population: All randomized participants in Part 1 who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 509 | 502
Participants | 475 | 453

8. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE is defined as "any untoward medical occurrence in a participant which does not necessarily have to have a causal relationship with this treatment". An AE can therefore be any unfavorable and unintended signs (such as rash or enlarged liver), symptoms (such as nausea or chest pain), an abnormal laboratory finding (including results of blood tests, x-rays or scans) or a disease temporarily associated with the use of the protocol treatment, whether or not considered related to the investigational medicinal product. The number of participants who discontinued study treatment due to an AE was reported for all participants in each treatment arm.
Time Frame: Up to 22 months
Population: All randomized participants in Part 1 who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 509 | 502
Participants | 70 | 18

9. Secondary Outcome: Clearance (CL) of Pembrolizumab
Description: Blood samples were to be collected at pre-specified time points and plasma isolated for analysis of pembrolizumab CL, defined as the volume of plasma from which pembrolizumab is eliminated per unit time following IV pembrolizumab administration. Samples were not collected and this analysis was not performed.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 4, 6, and 8, and then Day 1 of cycle for every 4 cycles afterwards (up to approximately 16 months). Each cycle is 3 weeks.
Population: As pre-specified by the protocol, pembrolizumab CL was not analyzed as planned and no data were collected since by the time of the interim analysis, pembrolizumab pharmacokinetics (PK) in melanoma patients had been well characterized and found to be consistent with the overall clinical pharmacology of pembrolizumab characterized across indications.
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Volume of Distribution (V) of Pembrolizumab
Description: Blood samples were to be collected at pre-specified time points and plasma isolated for analysis of pembrolizumab V, defined as the theoretical volume that would be necessary to contain the total amount of administered pembrolizumab at the same concentration that it is observed in the blood plasma. Samples were not collected and this analysis was not performed.
Time Frame: as for outcome 9
Population: As pre-specified by the protocol, pembrolizumab V was not analyzed as planned and no data were collected since by the time of the interim analysis, pembrolizumab PK in melanoma patients had been well characterized and found to be consistent with the overall clinical pharmacology of pembrolizumab characterized across indications.
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants Positive for Anti-Drug Antibodies (ADA) After Pembrolizumab Treatment
Description: Pre- and post-baseline serum samples from participants treated with pembrolizumab were analyzed for ADA by means of a neutralizing antibody assay which assessed the ability of ADA to block (neutralize) binding of pembrolizumab to Programmed Cell Death-1 (PD-1) protein. Overall immunogenicity was defined as the number of treatment emergent positive participants based on the total number of evaluable participants (treatment emergent positive, non-treatment emergent positive and negative immunogenicity status).
Time Frame: as for outcome 9
Population: All randomized participants in Part 1 who had at least one ADA sample available after treatment with pembrolizumab and who had treatment emergent positive, non-treatment emergent positive, or negative immunogenicity status. Participants receiving Placebo treatment in Part 1 were not analyzed for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Placebo
Number analyzed (Participants) | 495 | 0
Participants
  Negative | 473 |
  Non-Treatment emergent positive | 5 |
  Treatment emergent positive | 17 |

ADVERSE EVENTS:
Time Frame: Up to 29 months (through database cut-off date of 02-Oct-2017)
Description: All-Cause Mortality was reported for all randomized participants in Part 1.
  Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment in Part 1. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 25/514 | 35/505
Serious Adverse Events (participants affected / at risk) | 128/509 | 82/502
Other Adverse Events (participants affected / at risk) | 443/509 | 409/502
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=509) | Placebo (N=502)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune pericarditis (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 3 (3) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 2 (2) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aptyalism (Gastrointestinal disorders) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 3 (6) | 0 (0)
Colitis (Gastrointestinal disorders) | 8 (11) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (9) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (3)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral lichen planus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Papillitis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (8) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 2 (8) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Sarcoidosis (Immune system disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (4) | 7 (8)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 4 (4)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (4) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 (24) | 25 (36)
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leydig cell tumour of the testis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (4)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (10) | 3 (4)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (4)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=509) | Placebo (N=502)
Hyperthyroidism (Endocrine disorders) | 52 (61) | 6 (6)
Hypothyroidism (Endocrine disorders) | 75 (93) | 14 (14)
Abdominal pain (Gastrointestinal disorders) | 37 (40) | 31 (37)
Constipation (Gastrointestinal disorders) | 34 (37) | 29 (32)
Diarrhoea (Gastrointestinal disorders) | 140 (238) | 129 (234)
Dry mouth (Gastrointestinal disorders) | 30 (32) | 10 (10)
Nausea (Gastrointestinal disorders) | 88 (112) | 73 (103)
Vomiting (Gastrointestinal disorders) | 40 (55) | 22 (25)
Asthenia (General disorders) | 56 (93) | 42 (71)
Fatigue (General disorders) | 168 (247) | 168 (232)
Influenza like illness (General disorders) | 55 (73) | 38 (47)
Nasopharyngitis (Infections and infestations) | 44 (54) | 25 (26)
Upper respiratory tract infection (Infections and infestations) | 39 (49) | 30 (39)
Alanine aminotransferase increased (Investigations) | 35 (41) | 24 (30)
Weight decreased (Investigations) | 55 (69) | 39 (64)
Weight increased (Investigations) | 63 (96) | 82 (117)
Decreased appetite (Metabolism and nutrition disorders) | 36 (40) | 13 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 79 (130) | 72 (98)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (37) | 54 (69)
Myalgia (Musculoskeletal and connective tissue disorders) | 35 (40) | 25 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 (26) | 30 (34)
Dizziness (Nervous system disorders) | 26 (29) | 31 (38)
Headache (Nervous system disorders) | 95 (135) | 93 (126)
Cough (Respiratory, thoracic and mediastinal disorders) | 70 (88) | 55 (66)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 46 (50) | 25 (26)
Pruritus (Skin and subcutaneous tissue disorders) | 99 (138) | 58 (74)
Rash (Skin and subcutaneous tissue disorders) | 67 (90) | 43 (51)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27 (44) | 24 (26)
Hypertension (Vascular disorders) | 74 (178) | 77 (209)
Lymphoedema (Vascular disorders) | 26 (28) | 36 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All draft publications, including abstracts or detailed summaries of any proposed presentations, must be submitted to the Sponsor at the earliest practicable time for review, not less than 30 days before submission or presentation unless otherwise set forth in the clinical trial agreement. Sponsor shall have the right to delete any confidential information contained in any proposed presentation or abstract and may delay publication for up to 60 days for purposes of filing a patent application.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT02362594/Prot_SAP_000.pdf